CLINICAL TRIAL: NCT05200403
Title: Quantification of Improvement In Scratch Behavior And Sleep In Patients With Atopic Dermatitis on Crisaborole Ointment, 2%
Brief Title: Improvement In Scratch Behavior And Sleep In Patients With Atopic Dermatitis
Acronym: PAD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding was stoppped by grantor.
Sponsor: Boston University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-42240; H-42240 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
Keywords: Night-time itch; Night-time scratch; Crisaborole; Children 3 months to ≤ 11 years; Accelerometry; Actigraphy; Quality of life; Vehicle
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Crisaborole 2% (Experimental): Adult caregivers of children participants will be asked to apply a thin even-layer of Crisaborole (2%) twice daily for 2 weeks.
  Interventions: Drug: Crisaborole 2%; Device: Accelerometry device for children; Device: Accelerometry device for adult caregivers
- Vehicle Arm (Active Comparator): Adult caregivers of children participants will be asked to apply a thin even-layer of vehicle treatment twice daily for 2 weeks.
  Interventions: Drug: Vehicle treatment; Device: Accelerometry device for children; Device: Accelerometry device for adult caregivers

INTERVENTIONS:
Drug: Crisaborole 2% — The adult caregiver will apply a thin layer of Crisaborole 2% topically on their child participant twice a day for 2 weeks.
  Other Names: EUCRISA
  Arms: Crisaborole 2%
Drug: Vehicle treatment — The adult caregiver will apply a thin layer of the vehicle treatment topically on their child participant twice a day for 2 weeks. The vehicle treatment is made of excipients of crisaborole ointment (non-medicated ointment).
  Other Names: Nonmedicated ointment
  Arms: Vehicle Arm
Device: Accelerometry device for children — Children participants will wear two wrist worn (or wrist worn AND ankle worn for 3 months up to <2 years) accelerometry devices. Devices will be optional for child participants who have active AD on location of device placement, with a minimum of at least one wrist device needed for enrollment.
Device: Accelerometry device for adult caregivers — Adult caregiver participants will wear two accelerometry devices (one on each wrist) and complete daily assessments related to scratching, sleeping habits, pain, AD severity, quality of life, and device comfort questionnaires.

SUMMARY:
This single blind study is to primarily evaluate wearable devices and Observer Reported Itch Assessment in children to assess reduction of itch and night-time scratch in response to Crisaborole treatment vs. vehicle treatment (active control comparator without crisaborole) in children with atopic dermatitis (AD). Participants, age 3 months to 11 years with symptomatic mild to moderate AD, along with their primary caregivers will be recruited.

The goal of this study is to more fully evaluate the rapid onset of night-time itch and scratch relief, as well as improvements in sleep following treatment with Crisaborole in comparison to vehicle treatment in children with AD. the study will also assess the quality of life (QoL) and sleep within the associated caregivers.

DETAILED DESCRIPTION:
Approximately 270 children participants, age 3 months to ≤ 11 years, and their primary caregiver participants, for a total of 540 participants (270 pairs) will be randomized in 1:1 ratio to either Crisaborole (2% BID) or vehicle treatment and will be followed for 2 weeks. Participants will be asked to apply a thin even-layer of Crisaborole (2%) or vehicle twice daily (BID), excluding mouth, eyes, and vagina, per label, to all locations with active lesions (except for hands/fingers or within 1 to 2 fingers of the mouth to avoid inadvertent ingestion of ointment) and record location and time of application on the daily dosing form (provided by study staff, and as identified on the Dosing Record Sheet, breastfeeding women will be instructed to use the provided gloves when applying Crisaborole/vehicle). The study will be comprised of an initial screening/baseline visit for children participants who have an existing diagnosis of symptomatic AD, screened and enrolled in the study along with their primary caregivers after signing an informed consent (for parents/guardians and assent when appropriate).

Primary Objective:

1. Evaluate the effects of Crisaborole on itch and night-time scratch (as measured by accelerometry/actigraphy and Observer Reported Itch Assessment (3 months to ≤ 11 years old)) in children with mild to moderate AD between the ages of 3 months to ≤ 11 years old.

Secondary Objectives:

1. Evaluate the effects of Crisaborole on sleep in children ages 3 months to ≤ 11 years with mild to moderate AD.
2. Evaluate sleep in primary caregivers.
3. Evaluate the QoL measures in response to Crisaborole treatment (children 3 months to ≤ 11 years).
4. Evaluate QoL measures in response to the child's treatment, to the parents/caregivers/families.
5. Evaluate the effect of crisaborole treatment on AD signs, symptoms and severity in children ages 3 months to ≤ 11 years with mild to moderate AD.

The study will consist of a screening/baseline (in-laboratory) visit on Day -7 (V01), an in-laboratory visit Day 1 (V02), an in-laboratory visit on Day 2 (V03) for tape-striping, and Day 8 (V04) for a clinical assessment of the severity of the AD and a final in-laboratory visit on Day 15 (V05) for an assessment of the AD, tape-stripping, completion of ObsROs and return devices. Throughout the study, the participants and caregivers will wear accelerometry devices continuously (optional for those who have active AD on location of device placement, with a minimum of at least one wrist device needed for enrollment; devices may be removed for short periods of time for such things as the purposes of bathing, etc.). Enrolled participants will be randomly assigned to each arm of the study. Participants may come in for an unscheduled visit as needed (i.e., to replace compound, etc.). All in-person study activities, including informed consent and pregnancy testing, will be completed at the Laboratory for Human Neurobiology, 650 Albany St X140, Boston, MA, 02118. All activities performed in the laboratory are accomplished in private rooms. Primary caregivers will be provided with ample time and a privacy curtain to change into a gown during assessment for exclusion of Atopic Dermatitis, and primary caregivers will accompany children during all activities to ensure participant privacy. All at-home study activities will be completed in the participants' home.

ELIGIBILITY:
Inclusion Criteria for Children (3 months to ≤ 11 years):

1. Male or female participants aged between ≥3 months of age and ≤ 11 years of age at Day -7.
2. Written informed consent from participant/parent(s)/guardian(s).
3. Native English speakers or demonstrated fluency in English (as age appropriate).
4. Participants and parent(s)/guardian(s) are willing and able to comply with study instructions, study visits, procedures, and device placement (devices will be optional for those who have active AD on location of device placement, with a minimum of at least one wrist device needed for enrollment).
5. Have a clinical diagnosis of AD according to the criteria of Hanifin and Rajka.
6. Have AD involvement ≥ 5% Treatable % Body Surface Area (BSA) excluding the scalp and less than 40% BSA.
7. Have an Investigator's Static Global Assessment (ISGA) score of Mild (2) or Moderate (3) at the baseline visit.
8. Have an Eczema Area and Severity Index (EASI) total score of ≥3 at Day -7.
9. Have a minimum Observer Reported Itch Assessment score of 2 at Day -7 (ages 3 months - ≤ 5 years only) or a minimum Patient Reported Itch Severity Scale score of 2 (ages 6 years - ≤ 11 years old) at Day -7.
10. Participant/parent(s)/guardian(s) agrees to refrain from applying diaper rash creams, lotions, ointments, powders, etc. where AD lesions are present, unless AD lesions are present where crisaborole cannot be applied (face within 1 or 2 fingers away from the mouth and hands/fingers).
11. Participants must agree to refrain from applying crisaborole/vehicle to AD lesions on the fingers or hands or within 1 or 2 fingers away from the the mouth to prevent inadvertent ingestion of ointment.

Inclusion Criteria for Adult Caregiver (18-75 years):

1. Primary caregiver of the enrolled child participant, between ≥18 years of age and ≤75 years of age.
2. Able to understand and cooperate with study procedures and give informed consent.
3. Native English speakers or demonstrated fluency in English
4. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
5. ISGA score of 0 or 1 of AD at the screening visit, and no reported diagnosis of Atopic Dermatitis
6. WRAT-4 Word Reading Subtest equivalent to 8th grade reading level or greater.

Exclusion Criteria for Children:

1. Has any clinically significant medical disorder, condition, disease (including active or potentially recurrent non-AD dermatological conditions and known genetic dermatological conditions that overlap with AD, such as Netherton syndrome) or clinically significant finding at baseline that precludes participant's participation in study activities.
2. Participants who are on systemic corticosteroids or immunosuppressive agents within 28 days of Day -7 (V01).
3. 3. Participants who are on topical AD treatment such as low-to-high-potency corticosteroids, TCIs, antihistamines, antibiotics, sodium hypochlorite-based products, antibacterial soaps, bleach baths, diaper rash creams, lotions, ointments, powders, light therapy, and use of bland emollients on or overlapping with treatable AD-involved areas within 7 days of Day -7 (V01), unless AD lesions are present where crisaborole cannot be applied (face within 1 or 2 fingers away from the of mouth and hands/fingers).
4. Participants who are or have been on crisaborole treatment regimen in the past.
5. Allergy to polyurethane resin (strap/wristband component), skin nickel allergy, silicone, and/or adhesives.
6. Has documented non-AD related insomnia, sleep apnea or other sleep-related disorders (e.g., narcolepsy, restless legs syndrome, circadian rhythm disorder).
7. Participant has a known lack of efficacy to crisaborole.
8. Participant scores <20 on the Childhood Asthma Control Test (ages 4-≤ 11) indicating poorly controlled asthma.
9. If participant has a history of angioedema or anaphylaxis.
10. Has a significant active systemic or localized infection, including actively infected.
11. Has any planned surgical or medical procedure that would overlap with study participation.
12. Participants with cardiac pacemakers, electronic pumps or any other implanted medical devices.
13. Participants who are unable to wear at least one wrist device (one accelerometry device on at least one wrist).

Exclusion Criteria for Adult Caregiver:

1. Has any clinically significant medical disorder, condition, disease or clinically significant finding at screening that precludes Caregivers participation in study activities (e.g., sleep apnea, narcolepsy, etc.)
2. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1drink=5ounces (150mL) wine, 12 ounces (360mL) of beer, or 1.5 ounces (45mL) of hard liquor) within 6 months of screening as disclosed by participant during evaluation.
3. Current shift worker or travel across more than two time zones in the past 2 weeks, and/or during the study period.
4. Has any planned surgical or medical procedure that would overlap with study participation.
5. Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are Boston University (BU)/Boston Medical Center (BMC) employees directly involved in the conduct of the study.
6. Allergy to polyurethane resin (strap/wristband component), skin nickel allergy, silicone, and/or adhesives.
7. A female who is pregnant.
8. The primary caregiver or share the same domicile of another child who has previously been or is currently enrolled in the study.

Ages: 3 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Thomas, PhD, Principal Investigator — BU School of Medicine, Anatomy and Neurobiology
Locations (1):
- BU CAMed Laboratory for Human Neurobiology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Caregiver: Caregivers of Child Participants; caregivers did not receive treatment with crisaborole or vehicle.
Period: Overall Study
Arm/Group | Crisaborole 2% | Vehicle Arm | Caregiver
Started | 21 | 15 | 36
Completed | 17 | 13 | 30
Not Completed | 4 | 2 | 6
Not completed — Withdrawal by Subject | 4 | 2 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Crisaborole 2% | Vehicle Arm | Caregiver | Total
Number analyzed (Participants) | 21 | 15 | 36 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 15 | 0 | 36
  Between 18 and 65 years | 0 | 0 | 36 | 36
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 34 | 51
  Male | 10 | 9 | 2 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 9 | 19 | 40
  White | 5 | 4 | 10 | 19
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 1 | 1 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 21 | 15 | 36 | 72
Observer Reported Itch Assessment (ORIA) [Mean (Standard Deviation); unit: score on a scale] — Observer Reported Itch Assessment (ORIA) as recorded at participant intake. The ORIA is an 11 point likert scale that determines the caregiver's observation of the child's itch at the worst moment during the previous 24 hours with 0 being "No itch" and 10 being "Worst Itch Imaginable." The caregiver does not answer the ORIA about their own itch, only their child's itch, therefore, Observer Reported Itch Assessment data were not collected for the Caregiver Arm/Group. Population: Observer Reported Itch Assessment were not collected for Caregiver Arm/Group.
  score on a scale
    number analyzed (Participants) | 21 | 15 | 0 | 36
    (all) | 5.48 (2.09) | 6.61 (2.31) |  | 6.07 (2.30)
Number of children's nighttime scratching episodes [Mean (Standard Deviation); unit: scratch count per night] — The number of nighttime scratching episodes recorded by accelerometry. Population: For the crisaborole group, there were 11 participants that had sufficient processable data. For the Vehicle group, there were 8 participants that had sufficient processable data. The rest were not included due to device malfunction, non-wear, or missing data. The number of children's nighttime scratching episodes were not collected for the Caregiver Arm/Group.
  scratch count per night
    number analyzed (Participants) | 11 | 8 | 0 | 19
    (all) | 104.83 (54.49) | 103.82 (69.22) |  | 104.33 (61.86)
Duration of children's nighttime scratching episodes [Mean (Standard Deviation); unit: minutes] — The duration of nighttime scratching episodes recoded by accelerometry. Population: For the crisaborole group, there were 11 participants that had sufficient processable data. For the Vehicle group, there were 8 participants that had sufficient processable data. The rest were not included due to device malfunction, non-wear, or missing data. The duration of children's nighttime scratching episodes were not collected for the Caregiver Arm/Group.
  minutes
    number analyzed (Participants) | 11 | 8 | 0 | 19
    (all) | 7.81 (4.33) | 7.44 (5.50) |  | 7.63 (4.92)

OUTCOME MEASURES:

1. Primary Outcome: Number of Children's Nighttime Scratching Episodes
Description: The number of nighttime scratching episodes will be recorded on by accelerometry.
Time Frame: 2 weeks
Population: For the crisaborole group, there were 11 participants that had sufficient processable data. For the Vehicle group, there were 8 participants that had sufficient processable data. The rest were not included due to device malfunction, non-wear, or missing data.
Measure: Mean (Standard Deviation); unit: scratch count per night
Arm/Group | Crisaborole 2% | Vehicle Arm
Number analyzed (Participants) | 11 | 8
scratch count per night | 93.04 (70.35) | 116.85 (62.17)

2. Primary Outcome: Duration of Children's Nighttime Scratching Episodes
Description: The duration of nighttime scratching episodes will be recorded on by accelerometry.
Time Frame: 2 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Crisaborole 2% | Vehicle Arm
Number analyzed (Participants) | 11 | 8
minutes | 7.04 (6.44) | 8.63 (5.00)

3. Primary Outcome: Scratch Assessment by Adult Caregiver
Description: Adult caregivers will fill out the Observer Reported Itch Assessment (ORIA) which is a single question assessment to assess the severity of the child participant's itch. The minimum score of "0" indicates "no itch" and the maximum score of "10" indicates "worst itch imaginable."
Time Frame: 2 weeks
Population: 1 participant from each group withdrew after visit 1, thus no at home data was collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crisaborole 2% | Vehicle Arm
Number analyzed (Participants) | 20 | 14
score on a scale | 3.91 (2.45) | 3.53 (2.05)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Crisaborole 2% | Vehicle Arm | Caregiver
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/15 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/15 | 0/36
Other Adverse Events (participants affected / at risk) | 1/21 | 0/15 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crisaborole 2% (N=21) | Vehicle Arm (N=15) | Caregiver (N=36)
Overall Study (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Atopic Dermatitis flare up in the location of wearable sensors on both wrists. Adverse Events were assessed systematically based on routine monitoring during in-laboratory visits, which is where this event was discovered.

LIMITATIONS AND CAVEATS:
Funding was stopped by grantor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT05200403/Prot_SAP_000.pdf